CLINICAL TRIAL: NCT01544790
Title: Robot-assisted Minimally Invasive Thoraco-laparoscopic Esophagectomy Versus Open Transthoracic Esophagectomy for Resectable Esophageal Cancer. The ROBOT-trial: a Monocenter Randomized Controlled Trial.
Brief Title: Robot-assisted Thoraco-laparoscopic Esophagectomy Versus Open Transthoracic Esophagectomy
Acronym: ROBOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Richard van Hillegersberg, Prof., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL35048.041.11; 11141 (Registry Identifier: NTR3291)
Record Dates: First submitted 2012-02-17; First posted 2012-03-06 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Carcinoma; Esophageal Cancer
Keywords: Esophageal carcinoma; Esophageal cancer; Robotic surgery; Esophagectomy; Minimally invasive
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot-assisted esophagectomy (Experimental): Robot-assisted thoraco-laparoscopic esophagectomy with gastric conduit formation.
  Interventions: Procedure: Esophagectomy
- Open transthoracic esophagectomy (Active Comparator): traditional open transthoracic esophagectomy with gastric conduit formation.
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — In this monocenter prospective randomized controlled trial, we compare robot-assisted minimally invasive esophagectomy with conventional open transthoracic esophagectomy.
  Other Names: robot-assisted minimally invasive esophagectomy; robot-assisted thoraco-laparoscopic esophagectomy

SUMMARY:
This is the first randomized controlled trial designed to compare robot-assisted minimally invasive thoraco-laparoscopic esophagectomy with open transthoracic esophagectomy as surgical treatment for resectable esophageal cancer.

If our hypothesis is proved correct, robot-assisted minimally invasive thoraco-laparoscopic esophagectomy will result in a lower percentage of postoperative complications, lower blood loss, shorter hospital stay, but with at least similar oncologic outcomes and better postoperative quality of life compared with the open transthoracic esophagectomy (current standard).

DETAILED DESCRIPTION:
Rationale: As stated in the 2010 revised Dutch esophageal carcinoma guidelines, the golden standard for surgical treatment of esophageal carcinoma is open transthoracic esophagectomy. Recent evidence suggests that robot-assisted thoraco-laparoscopic esophagectomy using the Da Vinci ® robot can provide an extensive resection, with possibly better or at least equal radical (R0) resection rates and an equal number of dissected lymph nodes. This is accompanied with markedly reduced blood loss and reduction of overall complications with shorter intensive care unit (ICU) and hospital stay. Therefore, the robot-assisted thoraco-laparoscopic esophagectomy is now at a stage that it should be compared to the current standard of care in a randomized controlled trial.

Objective: Evaluate the benefits, risks and costs of robot-assisted thoraco-laparoscopic esophagectomy as an alternative to open transthoracic esophagectomy as treatment for esophageal cancer.

Study design: Randomized controlled parallel-group superiority trial Study population: Patients (age ≥ 18 and ≤ 75 jaar) with histologically proven surgically resectable (cT1-4a, N0-3, M0) squamous cell carcinoma, adenocarcinoma or undifferentiated esophageal carcinoma of the intrathoracic esophagus with European Clinical Oncology Group (ECOG) status 0, 1 or 2.

Intervention: 112 patients will be randomly allocated to either A) robot-assisted thoraco-laparoscopic esophagectomy (n=56) or B) open transthoracic esophagectomy (n=56).

Patients will receive the following interventions:

Group A. Robot-assisted thoraco-laparoscopic esophagectomy, with gastric conduit formation.

Group B. Open transthoracic esophagectomy, with gastric conduit formation.

Main study parameters/endpoints: Primary outcome is the percentage of overall complications (Grade 2 and higher) as stated by the modified Clavien-Dindo classification (MCDC).

Secondary outcomes are individual components of the primary endpoint (major and minor complications), (in hospital) mortality within 30 and 60 days, R0 resections, operation related events, postoperative recovery, oncologic outcomes, cost-effectiveness and quality of life.

Follow-up: 60 months after randomization

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma of the intrathoracic esophagus.
* Surgical resectable (T1-4a, N0-3, M0)
* Age ≥ 18 and ≤ 75 years
* European Clinical Oncology Group (ECOG) performance status 0,1 or 2
* Written informed consent

Exclusion Criteria:

* Carcinoma of the cervical esophagus
* Carcinoma of the gastro-esophageal junction (GEJ) with major tumor in the gastric cardia (Siewert III)
* Prior thoracic surgery at the right hemithorax or thorax trauma (rationale: these patients will undergo open resection)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Postoperative complications modified Clavien-Dindo classification (MCDC) grade 2 and higher | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The primary outcome of this study is the percentage of overall complications (Grade 2 and higher) as stated by the modified Clavien-Dindo classification of surgical complications (MCDC)

SECONDARY OUTCOMES:
Individual components of the primary endpoint (major and minor complications) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Major complications (MCDC grade 2-4) Including: myocardial infarction, anastomotic leakage (clinical or radiologic diagnosis), anastomotic stenosis, chylothorax (chylous leakage, presence of chylous in chest tubes or indication start medium chain triglycerides containing tube feeding (Vivonex®), gastric tube necrosis (proven by gastroscopy), pulmonary embolus, deep vein thrombosis, vocal cord palsy or paralysis.
  Minor complications (MCDC grade 1) Including: wound infections, pleural effusions, delayed gastric emptying
(In hospital) Mortality within 30 and 60 days | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks and within 30 days or 60 days
  (In hospital) mortality and mortality within 30 and 60 days will be reported. The cause of death and the results of the autopsy report will be noted.
R0 resections (%) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The pathological analysis will be finished within 2 weeks.
Operation related events | Day of surgery, up to 24 hours after surgery.
  Operation time is defined as time from incision until closure (minutes) for both the thoracic and the abdominal phase of the procedure. For the robotic procedure, set up time will be recorded separately. Unexpected events and complications occurring during the operation will be recorded (e.g. massive hemorrhage, perforation of other organs).
  Blood loss during operation (ml, per phase). In case of conversion to thoracotomy or laparotomy the reason for conversion has to be explained (absolute numbers/percentage).
Postoperative recovery | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Pain: Type and dose of used analgesics will be noted during the hospital admission period.
  Visual Analogue Scale (VAS) for pain will be noted at following times: pre-operatively and the first 10 days after surgery and a fixed periods during follow up (6 weeks, 6 months and yearly post-operatively up to 5 years).
  Length of intensive care unit (ICU) - medium care unit (MCU) stay (days). Length of hospital stay (days).
Oncologic outcomes | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months after surgery.
  2, 3 and 5 year disease free and overall survival
Quality of life | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months after surgery.
  Questionnaires will be required at following times:
  SF-36, EORTC QLQ-C30 (Dutch), EORTC OES18 (Dutch) and EQ-5D (Appendix 1 & 2) pre-operative < 5 days and 6 weeks, 6 months and yearly up to 5 years post-operatively.
Costs (euro) | 5 years follow up
  Direct general costs, due to extra operating room time and extra instruments. Indirect costs, such as reduced ICU or hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. van Hillegersberg, MD,PhD, Principal Investigator — UMC Utrecht, dept. of Surgery
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Sluis PC, van der Horst S, May AM, Schippers C, Brosens LAA, Joore HCA, Kroese CC, Haj Mohammad N, Mook S, Vleggaar FP, Borel Rinkes IHM, Ruurda JP, van Hillegersberg R. Robot-assisted Minimally Invasive Thoracolaparoscopic Esophagectomy Versus Open Transthoracic Esophagectomy for Resectable Esophageal Cancer: A Randomized Controlled Trial. Ann Surg. 2019 Apr;269(4):621-630. doi: 10.1097/SLA.0000000000003031. PMID 30308612
- [Derived] van der Sluis PC, Ruurda JP, van der Horst S, Verhage RJ, Besselink MG, Prins MJ, Haverkamp L, Schippers C, Rinkes IH, Joore HC, Ten Kate FJ, Koffijberg H, Kroese CC, van Leeuwen MS, Lolkema MP, Reerink O, Schipper ME, Steenhagen E, Vleggaar FP, Voest EE, Siersema PD, van Hillegersberg R. Robot-assisted minimally invasive thoraco-laparoscopic esophagectomy versus open transthoracic esophagectomy for resectable esophageal cancer, a randomized controlled trial (ROBOT trial). Trials. 2012 Nov 30;13:230. doi: 10.1186/1745-6215-13-230. PMID 23199187